CLINICAL TRIAL: NCT00041457
Title: Epidemiology of Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert James Glynn, PhD, Biostatistician; Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 1183
Record Dates: First submitted 2002-07-08; First posted 2002-07-09 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Cardiovascular Diseases; Thromboembolism; Peripheral Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Thromboembolism; Peripheral Vascular Diseases

GROUPS / COHORTS (4):
- Physicians' Health Study I
- Physicians' Health Study II
- Women's Health Study
- Women's Antioxidant Cardiovascular Health Study

SUMMARY:
To evaluate potentially modifiable lifestyle predictors of venous thromboembolism and their joint associations with biochemical and genetic determinants.

DETAILED DESCRIPTION:
BACKGROUND:

Venous thromboembolism is a common condition with considerable morbidity and mortality. The disorder has diverse causes including trauma, stasis, drugs, cancer, and genetic factors that contribute to enhanced clotting and coagulation. The study uses existing large-scale population studies to unravel factors responsible for and contributing to venous thromboembolism.

DESIGN NARRATIVE:

The study design is a prospective cohort study of 77,118 persons based on pooling information from four large randomized trials of US health professionals that have collected detailed risk factor information and have used common strategies to prospectively identify and validate cases of venous thromboembolism (VTE). These trials are: Physicians' Health Studies I & II including 29,071 US male physicians, of whom 22,071 have been followed since the initiation of the first trial in 1982; the Women's Health Study including 39,876 female health professionals who will have an average of 10 years of follow-up; and the Women's Antioxidant Cardiovascular Study including 8,171 female health professionals with prevalent cardiovascular disease or at high risk of cardiovascular disease who will have an average of 8 years of follow-up. Archived blood samples were collected from approximately 75 percent of participants at baseline and will be used to assess biochemical and genetic markers of risk including factor V Leiden, the G20210A mutation in the prothrombin gene, hyperhomocysteinemia, and anticardiolipin antibodies. The study will assess the joint association with risk of these markers and potentially modifiable factors including body mass index, hormone replacement therapy, physical activity, and aspirin use. The study population will include over 1,000 incident cases of VTE, including 750 with blood samples.

ELIGIBILITY:
No human subjects are involved. Collected data are used.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Glynn — Brigham and Women's Hospital

REFERENCES:
- [Background] Ridker PM, Goldhaber SZ, Danielson E, Rosenberg Y, Eby CS, Deitcher SR, Cushman M, Moll S, Kessler CM, Elliott CG, Paulson R, Wong T, Bauer KA, Schwartz BA, Miletich JP, Bounameaux H, Glynn RJ; PREVENT Investigators. Long-term, low-intensity warfarin therapy for the prevention of recurrent venous thromboembolism. N Engl J Med. 2003 Apr 10;348(15):1425-34. doi: 10.1056/NEJMoa035029. Epub 2003 Feb 24. PMID 12601075
- [Background] Glynn RJ, Rosner B. Comparison of risk factors for the competing risks of coronary heart disease, stroke, and venous thromboembolism. Am J Epidemiol. 2005 Nov 15;162(10):975-82. doi: 10.1093/aje/kwi309. Epub 2005 Oct 5. PMID 16207808